CLINICAL TRIAL: NCT02188082
Title: Clinical Trial of Systolic Heart Failure Treatment of IvabRadine Hemisulfate Sustained-release Tablets （FIRST）
Acronym: FIRST
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSQYFBLDHF2013
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Systolic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IvabRadine hemisulfate Sustained-release Tablets (Experimental): 5-15mg qd
  Interventions: Drug: IvabRadine hemisulfate Sustained-release Tablets
- placebo (Placebo Comparator): 5-15mg qd
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IvabRadine hemisulfate Sustained-release Tablets
  Arms: IvabRadine hemisulfate Sustained-release Tablets
Drug: placebo
  Arms: placebo

SUMMARY:
Ivabradine acts by inhibiting the ionic If current that modulates the pacemaker activity of sinoatrial node cells. The aim of present study is to evaluate the efficacy and safety of IvabRadine hemisulfate Sustained-release Tablets versus placebo in patients with moderate to severe chronic systolic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 75 years, males or females
* Willing to provide written informed consent
* NYHA Class II, III, or IV for≥4 weeks, in stable clinical condition for

  ≥4 weeks
* Optimized and unchanged chronic heart failure medications and dosages for≥4 weeks
* Sinus rhythm with resting heart rate≥70 b.p.m.
* Left-ventricular systolic dysfunction, with ejection fraction≥40% documented within previous 1 month

Exclusion Criteria:

* Unstable cardiovascular condition(for example, hospital admission for worsening heart failure)
* Recent (<2 months) myocardial infarction or recent or scheduled coronary revascularization
* Stroke or transient cerebral ischaemia within previous 4 weeks
* Severe primary valvular disease
* Scheduled surgery of valvular heart disease
* Active myocarditis
* Congenital heart diseases
* peripartum cardiomyopathy
* hyperthyroid heart disease
* On list for cardiac transplantation
* Cardiac resynchronization therapy started within previous 6 months
* Pacemaker with atrial or ventricular pacing (except biventricular pacing)˃40% of the time, or with stimulation threshold at the atrial or ventricular level˃60 b.p.m.
* Permanent atrial fibrillation or flutter
* Sick sinus syndrome, sinoatrial block, second and third degree atrio-ventricular block
* History of symptomatic or sustained (≥30 s) ventricular arrhythmia unless a cardioverter/defibrillator implanted
* Cardioverter/defibrillator shock within previous 6 months
* Family history or congenital long QT syndrome or treated with selected QT-prolonging products(except amiodarone)
* Contraindication or intolerance to ivabradine or lactulose
* Severe or uncontrolled hypertension (SBP≥180 mmHg or DBP≥110 mmHg)
* known anaemia(Hb<100 g/L)
* Known moderate or severe liver disease(ALT/AST˃3ULN), known severe renal disease(Cr˃2ULN)
* Pregnant or lactating women and women planning to become pregnant
* Use of an investigational drug within 30 days of enrollment
* Has a history of psychological illness/condition that interferes with ability to understand or complete requirements of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Left Ventricular End Systolic Volume Index by ultrasound cardiogram | baseline and week 32

SECONDARY OUTCOMES:
Change From Baseline in Left Ventricular End Diastolic Volume Index and left ventricular ejection fraction(LVEF) | baseline and week 32
incidence of hospital admission for worsening heart failure、any cardiovascular hospital admission、 cardiovascular mortality、all-cause mortality | baseline and week 32
change from baseline in distance of 6-minute walking test | baseline and week 32
change from baseline in heart rate | baseline and week 32
change from baseline in scores of Kansas City Cardiomyopathy Questionnaire | baseline and week 32
change from baseline in NT-proBNP | baseline and week 32

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (12):
- China (12):
  - The military general hospitla of Beijing PLA, Beijing, Beijing Municipality
  - The second affiliated hospital of suzhou university, Suzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - the First Hospital of Jilin University, Changchun, Jilin
  - shengjing hospital of China medical university, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - the Second Hospital of Shandong University, Jinan, Shandong
  - The first affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang
  - Hangzhou First People'S Hospital, Hangzhou, Zhejiang
  - The second affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang
  - The first affiliated hospital of wenzhou medical university, Wenzhou, Zhejiang
  - The second affiliated hospital of wenzhou medical university, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Ye F, Wang X, Wu S, Ma S, Zhang Y, Liu G, Liu K, Yang Z, Pang X, Xue L, Lu S, Zhong M, Li J, Yu H, Lou D, Cui D, Xie X, Wang J; FIRST Investigators. Sustained-Release Ivabradine Hemisulfate in Patients With Systolic Heart Failure. J Am Coll Cardiol. 2022 Aug 9;80(6):584-594. doi: 10.1016/j.jacc.2022.05.027. PMID 35926931